CLINICAL TRIAL: NCT00037934
Title: Evaluation of Robotic Upper Extremity Neuro-Rehabilitation
Brief Title: Robotic Upper-Limb Neurorehabilitation in Chronic Stroke Patient
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B2436
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Stroke
Keywords: Robot; Stroke; Upper Extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Robot exercise group
  Interventions: Device: Upper extremity robot
- 2 (Active Comparator): Traditional exercise group
  Interventions: Device: Upper extremity robot; Other: Traditional Supervised Upper Extremity Exercises

INTERVENTIONS:
Device: Upper extremity robot — Robotic upper extremity neuro-rehabilitation
Other: Traditional Supervised Upper Extremity Exercises — Arm ergometer, reaching, and stretching exercises
  Arms: 2

SUMMARY:
We have established the feasibility and effectiveness of robot-aided rehabilitation in stroke patients using a robot for neurological rehabilitation designed and built by MIT. Results of a pilot study of 20 patients were promising and showed that robot therapy is safe, tolerated by patients and produces a significant, measurable benefit. We propose to test that the robotic upper extremity trainer is an acceptable cost effective adjunct to standard occupational therapy for patients with dysfunction of the shoulder and elbow due to hemiparetic stroke in a VA rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Stroke
* Manual Muscle Score of Grade 3 or lower in at least one muscle of the affected arm

Exclusion Criteria:

* Acute Stroke
* Contracture or orthopedic problems limiting the movement of the affected arm
* Visual deficit such that the participant cannot see the test pattern on the robot trainer
* Serious complicating medical illness
* Botox treatment to the involved arm within three months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-04; Primary Completion 2004-09 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Upper limb Motor Status Score, Wolf Motor Function Test, Motor Power Assessment, and Fugl-Meyer Upper Extremity Motor Performance Test | The Primary Outcome measures were performed at baseline, after completion of 18 sessions of intervention and at 3 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bever, MD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States